CLINICAL TRIAL: NCT06419946
Title: Phase III Trial of Temozolomide/Lomustine (TMZ/LOM) Combination Therapy vs. Standard TMZ Therapy for Newly Diagnosed MGMT Promoter Methylated Glioblastoma (IDHwt) Patients +/- Tumor Treating Fields (Optune)
Brief Title: Lomustine in Addition to Standard of Care in Patients With MGMT Methylated Glioblastoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Skane University Hospital (Other); Gävle Hospital (Other); Karolinska Institutet (Other); Sahlgrenska University Hospital (Other); Karlstad Central Hospital (Other); Ryhov County Hospital (Other); Kalmar County Hospital (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); Sorlandet Hospital HF (Other Government); Helse Stavanger HF (Other Government); Aarhus University Hospital (Other); University Hospital, Umeå (Other); Eskilstuna Lasarettet (Other); Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506998-35-00
Record Dates: First submitted 2024-04-29; First posted 2024-05-17 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma, IDH-wildtype; MGMT-Methylated Glioblastoma
Keywords: precision medicine; temozolomide; lomustine; CCNU; survival
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Lomustine

STUDY DESIGN:
Intervention Model Description: Everyone: Radiotherapy (RT) consists of 60 Gy standard RT (RT 30x2Gy)
  Experimental treatment arm (TMZ/LOM):
  6 cycles of LOM/TMZ Start day 1 of RT. Cycle length of 42 days. Duration 9 months.
  Standard treatment arm (TMZ):
  Oral TMZ 75 mg/m2 daily during RT and with start day 1 of RT. This is followed by 6 cycles of TMZ with start 4 weeks after the end of RT. Cycle length 28 days. Duration 8,5 months.
  Everyone: TTFields start with radiotherapy/chemotherapy - but only in Sweden where TTF is part of standard of care (SOC). Ongoing until 2nd progression or max 2 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment arm (Experimental): arm with temozolomide (TMZ) plus lomustine (LOM) treatment.
  6 cycles of LOM/TMZ Start day 1 of RT. Cycle length of 42 days. Duration 9 months.
  Interventions: Drug: Temozolomide; Drug: Lomustine
- standard arm (Active Comparator): arm with standard of care treatment with temozolomide only.
  Oral TMZ 75 mg/m2 daily during RT and with start day 1 of RT. This is followed by 6 cycles of TMZ with start 4 weeks after the end of RT. Cycle length 28 days. Duration 8,5 months.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — In the experimental treatment arm: a combination of Temozolomide and Lomustine, taken together, two separate pills
  Other Names: TMZ
Drug: Lomustine — In the experimental treatment arm: a combination of Temozolomide and Lomustine, taken together, two separate pills
  Other Names: LOM
  Arms: treatment arm

SUMMARY:
Background: Glioblastoma (GBM) is notoriously difficult to treat, with current therapies often extending life by only a few months. The standard treatment involves surgery followed by radiation and chemotherapy with Temozolomide (TMZ). The efficacy of TMZ, however, is significantly enhanced when the tumor's o6-methylguanine-DNA-methyltransferase (MGMT) gene is methylated. Recent studies, such as the NOA-09 trial, have suggested that adding Lomustine (LOM) to TMZ could improve outcomes for patients with this specific tumor profile.

Hypothesis: The investigators hypothesize that the addition of LOM to the TMZ regimen will lead to significantly improved survival rates among patients with newly diagnosed glioblastoma who have a methylated MGMT promoter compared to those receiving only TMZ.

Treatment Plans: The study will randomly assign participants to two groups:

* Control Group: Standard treatment with TMZ during and after radiation therapy.
* Experimental Group: TMZ combined with LOM, starting on the first day of radiation therapy.

Outcome Measures: The primary outcome measure will be survival. Other outcomes will include progression-free survival (time from randomization until tumor progression or death), safety profiles (adverse effects of the treatments), and quality of life measures as well as neurocognitive outcomes.

DETAILED DESCRIPTION:
Current evidence:

In this section the investigators highlight the evidence behind the current standard fo care, and the emerging data supporting our approach. The RCT of Stupp showed that radiotherapy (RT) together with concomitant and adjuvant TMZ prolong survival. The NORDIC trial investigated the role of TMZ compared to RT for the subgroup of elderly patients, showing that survival was superior with TMZ, especially for those with mMGMT. LOM has been used for treatment of glioma for many decades, often used in combination with procarbazine and vincristine (PCV), but in recent years it is used in patients with glioblastoma as 2nd line therapy after failure of TMZ.

A phase 3 trial with Tumor Treating Fields (TTF, alternating low intensity electromagnetic fields) showed prolonged survival in patients with glioblastoma, but it is not universally applied/approved. Despite full multimodal treatment with surgery, RT, TMZ and TTFields, the median survival is <2 years. There is an unmet medical need to further improve treatments for these patients.

One RCT (NOA-09) provided preliminary data to exploit the specific vulnerability of mMGMT in glioblastoma (although no use of TTF in this trial). The overall tolerability of TMZ-LOM in combination was acceptable, as most adverse events (AE) were moderate and transient. Furthermore, health-related quality of life (HRQoL) and neurocognition did not differ between groups.

Estimated sample size and power:

Sample size calculation is based upon the results from the CeTeG/NOA-09 trial. Accounting for attrition, a total of 200 mMGMT GBM patients have to be randomised. Patients that drop-out before start of any therapy will be replaced, which will lead to more than 200 patients being randomized. For overall survival (OS) all patients that started day 1 of radiochemotherapy will be analysed (modified ITT). For per protocol all patients that have completed week 6 of treatment arm will be analysed for outcome. Patients lost to follow-up after the start of chemotherapy will be evaluated as observations censored at the time of dropout. Approximately 45% of newly diagnosed patients have a mMGMT, thus for 200 randomised patients a minimum of 445 patients will be screened.

Addition to the already described statistics:

Randomizations are stratified for center and for TTFields. The primary confirmatory analysis will be based on the modified intention-to-treat (mITT) population.

Survival parameters are measured in days starting from the day of randomization. Median time estimates as well as 95% confidence intervals will be reported. All additional analyses will be descriptive.

The statistical analysis plan (SAP) and blinding of statisticians will ensure analytic transparency and robustness.

Finally, similarly to avoid producing outdated results, the investigators plan to start TTF concomitant according to the Trident trial where results are expected soon. Nevertheless, if the Trident results are negative, the investigators will submit an amendment for using TTF according to the current standard of care. The reverse would not be possible in the middle of the trial as this has required extensive discussion, planning, and training with all sites. Balance with respect to TTF use is ensured with stratification in the randomization process.

Further details of study design of this phase 3, open-label, multicenter randomised controlled trial with parallel group design is presented under respective subheadings.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma/gliosarcoma, IDH wild type
* Methylated MGMT promoter
* World Health Organization performance status 0-2
* Age 18-70

Exclusion Criteria:

* Previous malignancy within 3 y or malignancy treated non-curatively
* Previous chemotherapy or radiotherapy involving the head
* Off-protocol tumor-specific treatment
* Serious comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2031-12-15 (Estimated)

PRIMARY OUTCOMES:
overall survival | Assessed from day of randomization to event or last day of follow-up (FU). Aanlyzed 36 months after last inclusion ensures that all patients have a potential of minimum 36 months FU
  visualized with Kaplan-Meier plot, tested with log-rank test

SECONDARY OUTCOMES:
progression free survival (PFS) | Assessed from day of randomization to event or last day of follow-up (FU). Aanlyzed 36 months after last inclusion ensures that all patients have a potential of minimum 36 months FU
  radiological or clinical PFS according to the modified Response Assessment in Neuro-Oncology (mRANO) criteria (Kaplan-Meier plot, log-rank test)
quality of life (QoL) | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  According to the EORTC Quality of Life Questionnaire (EORTC QLQ-30) with brain cancer module 20; Evaluate minimal clinically important difference (MCID) (i.e. clinically relevant difference) according to guidelines.
  These questionnaires contain a total of 30 + 20 QoL-related questions which are scored on a nominal scale (0-5 points); the result of each question is recorded for computerized examination and the questions relating to the same dimension of QoL (e.g. emotional well-being) are taken together for an overall score of this dimension. The scores for the different dimensions will be compared between repeated assessments throughout the trial and between the two arms of the trial.
  Analysed at 8 different time points:
  1. start of therapy = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
neurocognition - verbal memory | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Verbal Memory Test: Participants are tasked with learning and recalling 15 words. They are asked to recognize the words among 15 distractors (other words). The test is repeated at the end of the test session (after approximately 30 minutes). This test measures how well the participant can learn and recall words. Low scores indicate verbal memory difficulties.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - visual memory | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Visual Memory Test: Participants are tasked with learning and recalling 15 geometric shapes. They are asked to recognize these among 15 distractors (other shapes). The test is repeated at the end of the test session (after approximately 30 minutes). This test measures how well the participant can learn and recall geometric shapes. Low scores indicate visual memory difficulties.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs" (CNS = central nervous system), a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - motor speed and fine motor control | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Finger Tapping Test: The test measures motor speed and fine motor control. Participants are to perform three "tapping" sessions, lightly tapping the top of a key on the computer with each hand. This test measures how many "tappings" the participant performs with each hand. Motor speed varies according to hand dominance. Low scores indicate motor slowing.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - cognitive speed | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Symbol Digit Coding: The test measures cognitive speed during simultaneous cognitive processes such as visual scanning, visual perception, visual memory, and motor skills. Low scores may indicate impulsivity, perception difficulties, or impaired processing speed.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - simple and complex reaction time, inhibition/disinhibition, mental flexibility, and focused attention. | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Stroop Test: The test measures simple and complex reaction time, inhibition/disinhibition, mental flexibility, and focused attention. It also measures how well participants can adapt to changes and increasing complexity in the task. Long reaction times indicate mental slowing. A large number of errors indicate impulsivity, perception difficulties, or impaired processing speed.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - attention | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Attention Shift Test: The test measures how well participants can shift attention and perform simultaneous tasks. Participants must adjust their responses to temporarily changed rules. Normal/good scores are achieved with a high proportion of correct answers and short reaction times.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - attention, vigilance, and reaction time | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Continuous Performance Test: The test measures attention, vigilance, and reaction time. Most normal participants achieve nearly perfect results on this test. Long response times indicate mental slowing or impaired attention.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
neurocognition - Perception | done at baseline after informed consent, before randomisation and start of treatment, week 6 from start of treatment= end of radiotherapy, and every 24 weeks from start of treatment and for max 36 months.
  Emotional Perception Test: The test measures how well participants can perceive and identify specific emotions and their ability to perceive and understand social information. Low scores indicate difficulties with emotional perception.
  Analysed at 8 different time points:
  1. start of therapy (RT/chemotherapy/TTFields) = day 1
  2. since first assessment 6 weeks later: middle of the first months (1.5)
  3. from now on, every 6 months: month 7.5
  4. month 13.5
  5. month 19.5
  6. month 25.5
  7. month 31.5
  8. month 37.5 (end of the follow-up after 4 years)
  Patients will be monitored with the "CNS Vital Signs", a validated computerized test battery with proven sensitivity to detect cognitive impairments in patients with brain tumors. The battery consists of 8 subtests.
Adverse events (AE) | assessed from day of randomization to death or 36 months FU
  according to the Common Terminology Criteria for Adverse Events (CTCAE). (descriptive statistics between groups). A complementary analysis of AE by severity of event and by relationship to treatment will be performed (Chi2 test). Dose reductions, delay of therapy in subsequent courses and premature withdrawals will also be described.
  The Pharmacovigilance Sahlgrenska University Hospital will provide an unbiased evaluation of all serious adverse events. This ensures a qualified evaluation to support the sponsor to ensure patient safety. A Data Safety Monitoring Board (DSMB) is appointed to perform pre-planned interim analyses. Prompt ad-hoc meeting of the DSMB will be held in case of suspected unexpected serious adverse events. The committee can recommend a break or the stopping of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Annika Malmström, MD, PhD, Principal Investigator — University Hospital, Linkoeping

IPD SHARING:
Plan to Share IPD: Yes
Since the proposed randomized controlled trial (RCT) will be running for many year and since the investigators want to avoid outdated results, there will be - independent of the results of this proposed RCT - a collaboration to pool this study's data with the very similar phase 3 trial, the NOA-09 study. Here, the investigators will set a meta-analysis in place to balance clinical benefit with time and costs in a good manner. Hence, data is used for new sub-projects to endorse findings.

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Malmstrom A, Gronberg BH, Marosi C, Stupp R, Frappaz D, Schultz H, Abacioglu U, Tavelin B, Lhermitte B, Hegi ME, Rosell J, Henriksson R; Nordic Clinical Brain Tumour Study Group (NCBTSG). Temozolomide versus standard 6-week radiotherapy versus hypofractionated radiotherapy in patients older than 60 years with glioblastoma: the Nordic randomised, phase 3 trial. Lancet Oncol. 2012 Sep;13(9):916-26. doi: 10.1016/S1470-2045(12)70265-6. Epub 2012 Aug 8. PMID 22877848
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Weller M, Le Rhun E. How did lomustine become standard of care in recurrent glioblastoma? Cancer Treat Rev. 2020 Jul;87:102029. doi: 10.1016/j.ctrv.2020.102029. Epub 2020 May 4. PMID 32408220
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Herrlinger U, Tzaridis T, Mack F, Steinbach JP, Schlegel U, Sabel M, Hau P, Kortmann RD, Krex D, Grauer O, Goldbrunner R, Schnell O, Bahr O, Uhl M, Seidel C, Tabatabai G, Kowalski T, Ringel F, Schmidt-Graf F, Suchorska B, Brehmer S, Weyerbrock A, Renovanz M, Bullinger L, Galldiks N, Vajkoczy P, Misch M, Vatter H, Stuplich M, Schafer N, Kebir S, Weller J, Schaub C, Stummer W, Tonn JC, Simon M, Keil VC, Nelles M, Urbach H, Coenen M, Wick W, Weller M, Fimmers R, Schmid M, Hattingen E, Pietsch T, Coch C, Glas M; Neurooncology Working Group of the German Cancer Society. Lomustine-temozolomide combination therapy versus standard temozolomide therapy in patients with newly diagnosed glioblastoma with methylated MGMT promoter (CeTeG/NOA-09): a randomised, open-label, phase 3 trial. Lancet. 2019 Feb 16;393(10172):678-688. doi: 10.1016/S0140-6736(18)31791-4. Epub 2019 Feb 14. PMID 30782343
- [Background] Weller J, Tzaridis T, Mack F, Steinbach JP, Schlegel U, Hau P, Krex D, Grauer O, Goldbrunner R, Bahr O, Uhl M, Seidel C, Tabatabai G, Brehmer S, Bullinger L, Galldiks N, Schaub C, Kebir S, Stummer W, Simon M, Fimmers R, Coch C, Glas M, Herrlinger U, Schafer N. Health-related quality of life and neurocognitive functioning with lomustine-temozolomide versus temozolomide in patients with newly diagnosed, MGMT-methylated glioblastoma (CeTeG/NOA-09): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2019 Oct;20(10):1444-1453. doi: 10.1016/S1470-2045(19)30502-9. Epub 2019 Sep 2. PMID 31488360
- See also: PubMed ID: 15758009 — https://pubmed.ncbi.nlm.nih.gov/15758009/
- See also: PubMed ID: 22877848 — https://pubmed.ncbi.nlm.nih.gov/22877848/
- See also: PubMed ID: 15758010 — https://pubmed.ncbi.nlm.nih.gov/15758010/
- See also: PubMed ID: 32408220 — https://pubmed.ncbi.nlm.nih.gov/32408220/
- See also: PubMed ID: 29260225 — https://pubmed.ncbi.nlm.nih.gov/29260225/
- See also: PubMed ID: 30782343 — https://pubmed.ncbi.nlm.nih.gov/30782343/
- See also: PubMed ID: 31488360 — https://pubmed.ncbi.nlm.nih.gov/31488360/